CLINICAL TRIAL: NCT04426825
Title: A Single Arm, Phase II Study of Atezolizumab (MPDL3280A, Anti-PD-L1 Antibody) in Combination With Bevacizumab in Patients With EGFR Mutation Positive Stage IIIB-IV Non-Squamous Non-Small Cell Lung Cancer Pretreated With Epidermal Growth Factor Receptor Tyrosine-Kinase Inhibitors
Brief Title: A Study of Atezolizumab in Combination With Bevacizumab in Patients With EGFR Mutation Positive Stage IIIB-IV Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41256
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab plus Bevacizumab (Experimental): Participants will receive atezolizumab plus bevacizumab intravenously on Day 1 of each cycle. Treatment will continue until progressive disease, unacceptable toxicity, or death.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a dose of 1200 mg intravenously on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 mg/kg on Day 1 of each 21-day cycle.
  Other Names: Avastin

SUMMARY:
This is an open-label, single-arm, phase II, multicenter study designed to evaluated the efficacy and safety of atezolizumab in combination with bevacizumab in PD-L1-selected patients with Stage IIIB-IV Non-Squamous NSCLC harbored EGFR mutation after EGFR TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy ≥ 10 months
* Histologically or cytologically confirmed stage IIIB, IIIC, or IV non-squamous NSCLC. Patients with tumors of mixed histology are eligible if the major histological component appears to be non-squamous.
* No prior treatment for Stage IIIB, IIIC, or IV non-squamous NSCLC, with the following exceptions:

Patients with a sensitizing mutation in the EGFR gene must have experienced disease progression or were intolerant to treatment with one or more EGFR TKIs. Patients who have progressed on or were intolerant to first-line osimertinib or other thirdgeneration EGFR TKIs are eligible.

Patients who have progressed on or were intolerant to first- or second-generation EGFR TKIs, and who have no evidence of the EGFR T790M mutation after TKI therapy are eligible.

Patients who have progressed on or were intolerant to first- or second-generation EGFR TKIs and who have evidence of the T790M mutation must have also progressed on or were intolerant to osimertinib to be eligible.

* TKIs approved for treatment of NSCLC discontinued >7 days prior to enrollment.
* Measurable disease per RECIST v1.1. PD-L1 expression of ≥1% as documented through central testing of a representative tumor tissue specimen either from previously obtained archival tumor tissue or tissue obtained from a biopsy at screening
* ECOG Performance Status of 0-1
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases as determined by CT or MRI evaluation during screening and prior radiographic assessments
* History of leptomeningeal disease
* Prior chemotherapy or other systemic therapy for stage IIIB, IIIC, or IV disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* History of malignancy other than NSCLC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Current treatment with anti-viral therapy for HBV
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulations
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab, 6 months after the final dose of bevacizumab
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease within 6 months prior to initiation of study treatment
* History of Grade ≥ 2 hemoptysis within 1 month prior to enrollment
* Evidence of bleeding diathesis or coagulopathy. Current or recent use of aspirin, clopidogrel or treatment with dipyramidole, ticlopidine, or cilostazol
* Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to enrollment
* History of stroke or transient ischemic attack within 6 months prior to enrollment
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
* History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to enrollment
* History of intra-abdominal inflammatory process within 6 months prior to initiation of study treatment, including but not limited to active peptic ulcer disease, diverticulitis,or colitis
* Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Proteinuria
* Clear tumor infiltration into the thoracic great vessels is seen on imaging
* Clear cavitation of pulmonary lesions is seen on imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- China (10):
  - Beijing Cancer Hospital, Beijing
  - Beijing Hospital; Internal Medicine-Oncology, Beijing
  - Beijing Chest Hospital; Oncology Department, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital; Zhejiang Cancer Hospital cancer department, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Fang W, Fang J, Tian P, Fan Y, Yu Q, Zhang X, Wang Z, Liu X, Shi Y, Zhang L. Efficacy and Safety of Atezolizumab Plus Bevacizumab in Patients With Advanced NSCLC Who Received Pretreatment With EGFR-TKIs (ML41256): A Multicenter, Prospective, Single-Arm, Phase 2 Trial. Cancer Med. 2025 Dec;14(24):e71469. doi: 10.1002/cam4.71469. PMID 41388935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple investigational sites in China
Period: Overall Study
Arm/Group | Atezolizumab Plus Bevacizumab
Started | 23
Completed | 0
Not Completed | 23
Not completed — Death | 17
Not completed — Lost to Follow-up | 1
Not completed — Study terminated by sponsor | 5

BASELINE CHARACTERISTICS:
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Smoking History [Number; unit: Participants]
  Never | 16
  Current | 0
  Previous | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) was defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions >=4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).
Time Frame: Baseline up to approximately 10 months
Population: The evaluable population included all enrolled participants who received any amount of study treatment, had baseline and at least one post-baseline efficacy measurement.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 22
Percentage of Participants | 18.2 [5.19 to 40.28]

2. Secondary Outcome: Duration of Objective Response (DOR)
Description: Duration of objective response (DOR) was defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause whichever occurs first, as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline up to approximately 2.5 years
Population: The full analysis set (FAS) population included all enrolled participants who received any amount of at least one dose of any study treatment. The analysis population for this outcome measures included participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 4
Months | 6.36 [2.66 to NA] — NA = not estimable due to the limited number of events observed

3. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) was defined as the time from the start of the treatment to the first objective tumor response observed for participants who achieved CR or PR, as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline up to approximately 2.5 years
Population: The FAS population included all enrolled participants who received any amount of at least one dose of any study treatment. The analysis population for this outcome measures included participants with a confirmed response (CR or PR).
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 4
Months | 1.577 (0.490)

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) was defined as the proportion of participants who have a best overall response of CR or PR or stable disease (SD), as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline up to approximately 2.5 years
Population: The FAS population included all enrolled participants who received any amount of at least one dose of any study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Percentage of Participants | 65.2 [42.73 to 83.62]

5. Secondary Outcome: Overall Survival (OS)
Description: OS after enrollment was defined as the time from enrollment to death from any cause.
Time Frame: Baseline until death due to any cause (up to approximately 2.5 years)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Months | 14.06 [8.80 to 22.14]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline up to approximately 2.5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Months | 2.76 [1.35 to 4.07]

7. Secondary Outcome: PFS Rate at 6 and 12 Months
Description: PFS rate at 6 and 12 months is defined as the percentage of participants who have not experienced disease progression or death from any cause at 6 and 12 months, as determined by the investigator according to RECIST v1.1.
Time Frame: Baseline to 6 months and 12 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Percentage of participants
  6 months | 13.91 [3.49 to 31.36]
  12 months | 4.64 [0.33 to 19.26]

8. Secondary Outcome: OS Rate at 1 and 2 Years
Description: OS rate at 1 and 2 years was defined as the percentage of participants who have not experienced death from any cause at 1 and 2 years.
Time Frame: Baseline to 1 and 2 Years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Percentage of participants
  1 year | 52.17 [30.51 to 70.01]
  2 years | 30.43 [13.54 to 49.28]

9. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Percentage of participants with adverse events.
Time Frame: Baseline up to approximately 2.5 years
Population: The safety population is defined as all enrolled participants who received any amount of at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Participants | 23

10. Secondary Outcome: Percentage of Participants With Serious and Non-Serious Immune-Mediated Adverse Events (irAEs)
Description: Percentage of serious and non-serious immune-mediated adverse events related to atezolizumab treatment. The AESIs were graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria. The grading is as follows: Grade 1=Mild AE, Grade 2=Moderate AE, Grade 3=Severe AE, Grade 4=Life-threatening or disabling AE, Grade 5=Death related to AE.
Time Frame: Baseline up to approximately 2.5 years
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Participants
  Non-serious irAEs | 7
  Serious irAEs | 1

11. Secondary Outcome: Objective Response Rate (ORR) According to iRECIST
Description: Objective response rate (ORR) is defined as the proportion of participants with a complete response (CR) or partial response (PR) on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to Modified RECIST v1.1 (iRECIST).
Time Frame: Baseline up to approximately 2.5 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Percentage of Participants | 17.4 [4.95 to 38.78]

12. Secondary Outcome: Disease Control Rate (DCR) According to iRECIST
Description: Disease control rate (DCR) is defined as the proportion of participants who have a best overall response of CR or PR or stable disease (SD), as determined by the investigator according to modified RECIST v1.1 (iRECIST).
Time Frame: Baseline up to 2 years and approximately 5 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Percentage of Participants | 65.2 [42.73 to 83.62]

13. Secondary Outcome: Duration of Objective Response (DOR) According to iRECIST
Description: Duration of objective response (DOR) is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause whichever occurs first, as determined by the investigator according to modified RECIST v1.1 (iRECIST).
Time Frame: Baseline up to approximately 2.5 years
Population: The full analysis set (FAS) population included all enrolled participants who received any amount of at least one dose of any study treatment. The analysis population for this outcome measures included participants with a confirmed response (iCR or iPR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 4
Months | 6.36 [2.66 to NA] — NA = not estimable; could not be calculated due to too few events.

14. Secondary Outcome: Progression-Free Survival (PFS) According to iRECIST
Description: Progression-free survival (PFS) is defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by the investigator according to modified RECIST v1.1 (iRECIST).
Time Frame: Baseline up to approximately 2.5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Months | 2.76 [1.35 to 4.07]

15. Secondary Outcome: Progression-Free Survival (PFS) Rate at 12 Months According to iRECIST
Description: Progression-free survival (PFS) rate is defined as the time from enrollment to the first occurrence of disease progression or death from any cause, whichever occurs first at 12 months, as determined by the investigator according to modified RECIST v1.1 (iRECIST).
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Months | 4.64 [0.33 to 19.26]

16. Secondary Outcome: Time to Deterioation (TTD) Using EORTC
Description: Time to deterioration (TTD) using European Organization for Research and treatment of Cancer (EORTC) Quality-of-life Questionnaire Core 30 (QLQ C30) and its Lung Cancer Module (QLQ LC13) is defined as the time from baseline to the first time the patient's score shows a >=10 points increase above baseline in any of the following EORTC-transformed symptom subscale scores (whichever occurs first): cough, dyspnoea (single item), dyspnoea (multi-item subscale), chest pain, or arm/shoulder pain, whichever occurred first. Scores ranged from 0-10. A higher score represented more severe symptoms.
Time Frame: Baselsine up to approximately 1 year
Population: The FAS population included all enrolled participants who received any amount of at least one dose of any study treatment. The number of participants in the FAS with a non-missing baseline PRO assessment are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 22
Months
  Cough | NA [3.48 to NA] — NA = too few events to calculate the median and upper confidence interval (CI)
  Dyspnoea (single-item Q33) | NA [NA to NA] — NA = too few events to calculate the median, upper and lower CI
  Dyspnoea (single-item Q34) | NA [NA to NA] — NA = too few events to calculate the median, upper and lower CI
  Dyspnoea (single-item Q35) | NA [NA to NA] — NA = too few events to calculate the median, upper and lower CI
  Dyspnoea (multi-item) | NA [NA to NA] — NA = too few events to calculate the median, upper and lower CI
  Chest pain | NA [2.10 to NA] — NA = too few events to calculate the median, upper CI
  Arm/shoulder pain | NA [NA to NA] — NA = too few events to calculate the median, upper and lower CI

17. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) and Health Status
Description: The 30-item EORTC QLQ-C30 version 3 is composed by five multi-item function scales (physical, role, cognitive, emotional, and social), three multi-item symptom scales (fatigue, nausea and vomiting, and pain), six single-item symptom scales (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties), and a two-item global quality of life scale. All EORTC scales and single-item measures are linearly transformed so that each score has a range of 0-100. A high score for the functional and general health areas represent better functional status and quality of life. Higher scores for the symptom scales represent more symptoms or problems (poor quality of life). A participant was classified as improved if a decrement of 10 points or worse was observed in the change from baseline scores. A participant was classified as worsened if a 10-point or greater increase was observed in the change from baseline scores.
Time Frame: Baseline up to approximately 1 year
Population: The FAS population included all enrolled participants who received any amount of at least one dose of any study treatment. The number of participants in the FAS with a non-missing baseline PRO assessment are presented. As each participant had different treatment cycles, this resulted in different numbers of participants analyzed per cycle.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Units on a scale
  Global Quality of Life (QoL) - Baseline: number analyzed (Participants) | 22
  Global Quality of Life (QoL) - Baseline | 53.409 (28.132)
  Global QoL - Treatment Cycle 02: number analyzed (Participants) | 20
  Global QoL - Treatment Cycle 02 | 0.833 (28.855)
  Global QoL - Treatment Cycle 03: number analyzed (Participants) | 16
  Global QoL - Treatment Cycle 03 | -0.521 (27.465)
  Global QoL - Treatment Cycle 04: number analyzed (Participants) | 12
  Global QoL - Treatment Cycle 04 | -6.250 (28.007)
  Global QoL - Treatment Cycle 05: number analyzed (Participants) | 8
  Global QoL - Treatment Cycle 05 | -15.625 (24.975)
  Global QoL - Treatment Cycle 06: number analyzed (Participants) | 8
  Global QoL - Treatment Cycle 06 | -16.667 (23.987)
  Global QoL - Treatment Cycle 07: number analyzed (Participants) | 6
  Global QoL - Treatment Cycle 07 | -23.611 (20.012)
  Global QoL - Treatment Cycle 08: number analyzed (Participants) | 6
  Global QoL - Treatment Cycle 08 | -20.833 (43.381)
  Global QoL - Treatment Cycle 09: number analyzed (Participants) | 3
  Global QoL - Treatment Cycle 09 | -36.111 (4.811)
  Global QoL - Treatment Cycle 10: number analyzed (Participants) | 3
  Global QoL - Treatment Cycle 10 | -22.222 (19.245)
  Global QoL - Treatment Cycle 11: number analyzed (Participants) | 3
  Global QoL - Treatment Cycle 11 | -30.556 (4.811)
  Global QoL - Treatment Cycle 12: number analyzed (Participants) | 3
  Global QoL - Treatment Cycle 12 | -27.778 (9.623)
  Global QoL - Treatment Cycle 13: number analyzed (Participants) | 1
  Global QoL - Treatment Cycle 13 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Global QoL - Treatment Cycle 14: number analyzed (Participants) | 2
  Global QoL - Treatment Cycle 14 | -25.000 (11.785)
  Global QoL - Treatment Cycle 15: number analyzed (Participants) | 2
  Global QoL - Treatment Cycle 15 | -33.333 (0.000)
  Global QoL - Follow Up: number analyzed (Participants) | 1
  Global QoL - Follow Up | -16.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Global QoL - Follow Up 2: number analyzed (Participants) | 1
  Global QoL - Follow Up 2 | -16.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Global QoL - Follow Up 3: number analyzed (Participants) | 1
  Global QoL - Follow Up 3 | -25.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Physical Functioning - Baseline: number analyzed (Participants) | 22
  Physical Functioning - Baseline | 79.091 (15.437)
  Physical Functioning - Treatment Cycle 02: number analyzed (Participants) | 20
  Physical Functioning - Treatment Cycle 02 | -5.667 (20.207)
  Physical Functioning - Treatment Cycle 03: number analyzed (Participants) | 16
  Physical Functioning - Treatment Cycle 03 | -4.167 (15.490)
  Physical Functioning - Treatment Cycle 04: number analyzed (Participants) | 12
  Physical Functioning - Treatment Cycle 04 | -0.556 (11.177)
  Physical Functioning - Treatment Cycle 05: number analyzed (Participants) | 8
  Physical Functioning - Treatment Cycle 05 | -1.667 (14.584)
  Physical Functioning - Treatment Cycle 06: number analyzed (Participants) | 8
  Physical Functioning - Treatment Cycle 06 | -0.833 (10.947)
  Physical Functioning - Treatment Cycle 07: number analyzed (Participants) | 6
  Physical Functioning - Treatment Cycle 07 | -6.667 (10.328)
  Physical Functioning - Treatment Cycle 08: number analyzed (Participants) | 6
  Physical Functioning - Treatment Cycle 08 | -8.889 (10.037)
  Physical Functioning - Treatment Cycle 09: number analyzed (Participants) | 3
  Physical Functioning - Treatment Cycle 09 | -15.556 (16.777)
  Physical Functioning - Treatment Cycle 10: number analyzed (Participants) | 3
  Physical Functioning - Treatment Cycle 10 | -6.667 (6.667)
  Physical Functioning - Treatment Cycle 11: number analyzed (Participants) | 3
  Physical Functioning - Treatment Cycle 11 | -6.667 (6.667)
  Physical Functioning - Treatment Cycle 12: number analyzed (Participants) | 3
  Physical Functioning - Treatment Cycle 12 | -13.333 (17.638)
  Physical Functioning - Treatment Cycle 13: number analyzed (Participants) | 1
  Physical Functioning - Treatment Cycle 13 | -6.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Physical Functioning - Treatment Cycle 14: number analyzed (Participants) | 2
  Physical Functioning - Treatment Cycle 14 | -6.667 (9.428)
  Physical Functioning - Treatment Cycle 15: number analyzed (Participants) | 2
  Physical Functioning - Treatment Cycle 15 | 0.000 (0.000)
  Physical Functioning - Follow Up: number analyzed (Participants) | 1
  Physical Functioning - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Physical Functioning - Follow Up 2: number analyzed (Participants) | 1
  Physical Functioning - Follow Up 2 | 6.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Physical Functioning - Follow Up 3: number analyzed (Participants) | 1
  Physical Functioning - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Role Functioning - Baseline: number analyzed (Participants) | 22
  Role Functioning - Baseline | 81.061 (22.593)
  Role Functioning - Treatment Cycle 02: number analyzed (Participants) | 20
  Role Functioning - Treatment Cycle 02 | -7.500 (32.307)
  Role Functioning - Treatment Cycle 03: number analyzed (Participants) | 16
  Role Functioning - Treatment Cycle 03 | -7.292 (28.525)
  Role Functioning - Treatment Cycle 04: number analyzed (Participants) | 12
  Role Functioning - Treatment Cycle 04 | -4.167 (14.434)
  Role Functioning - Treatment Cycle 05: number analyzed (Participants) | 8
  Role Functioning - Treatment Cycle 05 | -4.167 (21.362)
  Role Functioning - Treatment Cycle 06: number analyzed (Participants) | 8
  Role Functioning - Treatment Cycle 06 | -4.167 (14.773)
  Role Functioning - Treatment Cycle 07: number analyzed (Participants) | 6
  Role Functioning - Treatment Cycle 07 | 0.000 (21.082)
  Role Functioning - Treatment Cycle 08: number analyzed (Participants) | 6
  Role Functioning - Treatment Cycle 08 | -8.333 (25.276)
  Role Functioning - Treatment Cycle 09: number analyzed (Participants) | 3
  Role Functioning - Treatment Cycle 09 | -11.111 (19.245)
  Role Functioning - Treatment Cycle 10: number analyzed (Participants) | 3
  Role Functioning - Treatment Cycle 10 | -11.111 (9.623)
  Role Functioning - Treatment Cycle 11: number analyzed (Participants) | 3
  Role Functioning - Treatment Cycle 11 | 0 (0)
  Role Functioning - Treatment Cycle 12: number analyzed (Participants) | 3
  Role Functioning - Treatment Cycle 12 | -5.556 (9.623)
  Role Functioning - Treatment Cycle 13: number analyzed (Participants) | 1
  Role Functioning - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Role Functioning - Treatment Cycle 14: number analyzed (Participants) | 2
  Role Functioning - Treatment Cycle 14 | 0.000 (0.000)
  Role Functioning - Treatment Cycle 15: number analyzed (Participants) | 2
  Role Functioning - Treatment Cycle 15 | 0.000 (0.000)
  Role Functioning - Follow Up: number analyzed (Participants) | 1
  Role Functioning - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Role Functioning - Follow Up 2: number analyzed (Participants) | 1
  Role Functioning - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Role Functioning - Follow Up 3: number analyzed (Participants) | 1
  Role Functioning - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Emotional Functioning - Baseline: number analyzed (Participants) | 22
  Emotional Functioning - Baseline | 76.894 (23.561)
  Emotional Functioning - Treatment Cycle 02: number analyzed (Participants) | 20
  Emotional Functioning - Treatment Cycle 02 | -2.083 (18.312)
  Emotional Functioning - Treatment Cycle 03: number analyzed (Participants) | 16
  Emotional Functioning - Treatment Cycle 03 | -0.521 (20.965)
  Emotional Functioning - Treatment Cycle 04: number analyzed (Participants) | 12
  Emotional Functioning - Treatment Cycle 04 | 0.000 (28.868)
  Emotional Functioning - Treatment Cycle 05: number analyzed (Participants) | 8
  Emotional Functioning - Treatment Cycle 05 | -5.208 (23.544)
  Emotional Functioning - Treatment Cycle 06: number analyzed (Participants) | 8
  Emotional Functioning - Treatment Cycle 06 | -4.167 (19.920)
  Emotional Functioning - Treatment Cycle 07: number analyzed (Participants) | 6
  Emotional Functioning - Treatment Cycle 07 | -12.500 (22.822)
  Emotional Functioning - Treatment Cycle 08: number analyzed (Participants) | 6
  Emotional Functioning - Treatment Cycle 08 | -8.333 (15.811)
  Emotional Functioning - Treatment Cycle 09: number analyzed (Participants) | 3
  Emotional Functioning - Treatment Cycle 09 | -13.889 (17.347)
  Emotional Functioning - Treatment Cycle 10: number analyzed (Participants) | 3
  Emotional Functioning - Treatment Cycle 10 | -16.667 (14.434)
  Emotional Functioning - Treatment Cycle 11: number analyzed (Participants) | 3
  Emotional Functioning - Treatment Cycle 11 | -19.444 (26.788)
  Emotional Functioning - Treatment Cycle 12: number analyzed (Participants) | 3
  Emotional Functioning - Treatment Cycle 12 | -2.778 (12.729)
  Emotional Functioning - Treatment Cycle 13: number analyzed (Participants) | 1
  Emotional Functioning - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Emotional Functioning - Treatment Cycle 14: number analyzed (Participants) | 2
  Emotional Functioning - Treatment Cycle 14 | 4.167 (5.893)
  Emotional Functioning - Treatment Cycle 15: number analyzed (Participants) | 2
  Emotional Functioning - Treatment Cycle 15 | 4.167 (5.893)
  Emotional Functioning - Follow Up: number analyzed (Participants) | 1
  Emotional Functioning - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Emotional Functioning - Follow Up 2: number analyzed (Participants) | 1
  Emotional Functioning - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Emotional Functioning - Follow Up 3: number analyzed (Participants) | 1
  Emotional Functioning - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Cognitive Functioning - Baseline: number analyzed (Participants) | 22
  Cognitive Functioning - Baseline | 79.545 (17.006)
  Cognitive Functioning - Treatment Cycle 02: number analyzed (Participants) | 20
  Cognitive Functioning - Treatment Cycle 02 | 1.667 (17.014)
  Cognitive Functioning - Treatment Cycle 03: number analyzed (Participants) | 16
  Cognitive Functioning - Treatment Cycle 03 | -2.083 (14.751)
  Cognitive Functioning - Treatment Cycle 04: number analyzed (Participants) | 12
  Cognitive Functioning - Treatment Cycle 04 | 1.389 (15.006)
  Cognitive Functioning - Treatment Cycle 05: number analyzed (Participants) | 8
  Cognitive Functioning - Treatment Cycle 05 | -8.333 (17.817)
  Cognitive Functioning - Treatment Cycle 06: number analyzed (Participants) | 8
  Cognitive Functioning - Treatment Cycle 06 | 2.083 (13.909)
  Cognitive Functioning - Treatment Cycle 07: number analyzed (Participants) | 6
  Cognitive Functioning - Treatment Cycle 07 | -16.667 (25.820)
  Cognitive Functioning - Treatment Cycle 08: number analyzed (Participants) | 6
  Cognitive Functioning - Treatment Cycle 08 | -11.111 (17.213)
  Cognitive Functioning - Treatment Cycle 09: number analyzed (Participants) | 3
  Cognitive Functioning - Treatment Cycle 09 | -5.556 (9.623)
  Cognitive Functioning - Treatment Cycle 10: number analyzed (Participants) | 3
  Cognitive Functioning - Treatment Cycle 10 | 5.556 (9.623)
  Cognitive Functioning - Treatment Cycle 11: number analyzed (Participants) | 3
  Cognitive Functioning - Treatment Cycle 11 | 0.000 (0.000)
  Cognitive Functioning - Treatment Cycle 12: number analyzed (Participants) | 3
  Cognitive Functioning - Treatment Cycle 12 | -5.556 (9.623)
  Cognitive Functioning - Treatment Cycle 13: number analyzed (Participants) | 1
  Cognitive Functioning - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Cognitive Functioning - Treatment Cycle 14: number analyzed (Participants) | 2
  Cognitive Functioning - Treatment Cycle 14 | 0.000 (0.000)
  Cognitive Functioning - Treatment Cycle 15: number analyzed (Participants) | 2
  Cognitive Functioning - Treatment Cycle 15 | -8.333 (11.785)
  Cognitive Functioning - Follow Up: number analyzed (Participants) | 1
  Cognitive Functioning - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Cognitive Functioning - Follow Up 2: number analyzed (Participants) | 1
  Cognitive Functioning - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Cognitive Functioning - Follow Up 3: number analyzed (Participants) | 1
  Cognitive Functioning - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Social Functioning - Baseline: number analyzed (Participants) | 22
  Social Functioning - Baseline | 67.424 (28.857)
  Social Functioning - Treatment Cycle 02: number analyzed (Participants) | 20
  Social Functioning - Treatment Cycle 02 | -3.333 (30.874)
  Social Functioning - Treatment Cycle 03: number analyzed (Participants) | 16
  Social Functioning - Treatment Cycle 03 | 1.042 (25.436)
  Social Functioning - Treatment Cycle 04: number analyzed (Participants) | 12
  Social Functioning - Treatment Cycle 04 | -1.389 (28.831)
  Social Functioning - Treatment Cycle 05: number analyzed (Participants) | 8
  Social Functioning - Treatment Cycle 05 | 0.000 (34.503)
  Social Functioning - Treatment Cycle 06: number analyzed (Participants) | 8
  Social Functioning - Treatment Cycle 06 | 2.083 (32.657)
  Social Functioning - Treatment Cycle 07: number analyzed (Participants) | 6
  Social Functioning - Treatment Cycle 07 | -13.889 (24.553)
  Social Functioning - Treatment Cycle 08: number analyzed (Participants) | 6
  Social Functioning - Treatment Cycle 08 | -11.111 (25.092)
  Social Functioning - Treatment Cycle 09: number analyzed (Participants) | 3
  Social Functioning - Treatment Cycle 09 | -11.111 (25.459)
  Social Functioning - Treatment Cycle 10: number analyzed (Participants) | 3
  Social Functioning - Treatment Cycle 10 | -11.111 (9.623)
  Social Functioning - Treatment Cycle 11: number analyzed (Participants) | 3
  Social Functioning - Treatment Cycle 11 | -11.111 (9.623)
  Social Functioning - Treatment Cycle 12: number analyzed (Participants) | 3
  Social Functioning - Treatment Cycle 12 | -5.556 (19.245)
  Social Functioning - Treatment Cycle 13: number analyzed (Participants) | 1
  Social Functioning - Treatment Cycle 13 | 16.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Social Functioning - Treatment Cycle 14: number analyzed (Participants) | 2
  Social Functioning - Treatment Cycle 14 | -8.333 (35.355)
  Social Functioning - Treatment Cycle 15: number analyzed (Participants) | 2
  Social Functioning - Treatment Cycle 15 | -8.333 (35.355)
  Social Functioning - Follow Up: number analyzed (Participants) | 1
  Social Functioning - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Social Functioning - Follow Up 2: number analyzed (Participants) | 1
  Social Functioning - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Social Functioning - Follow Up 3: number analyzed (Participants) | 1
  Social Functioning - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Fatigue - Baseline: number analyzed (Participants) | 22
  Fatigue - Baseline | 34.343 (22.979)
  Fatigue - Treatment Cycle 02: number analyzed (Participants) | 20
  Fatigue - Treatment Cycle 02 | 3.889 (25.814)
  Fatigue - Treatment Cycle 03: number analyzed (Participants) | 16
  Fatigue - Treatment Cycle 03 | 8.333 (20.488)
  Fatigue - Treatment Cycle 04: number analyzed (Participants) | 12
  Fatigue - Treatment Cycle 04 | 5.556 (24.845)
  Fatigue - Treatment Cycle 05: number analyzed (Participants) | 8
  Fatigue - Treatment Cycle 05 | 8.333 (17.568)
  Fatigue - Treatment Cycle 06: number analyzed (Participants) | 8
  Fatigue - Treatment Cycle 06 | 9.722 (13.849)
  Fatigue - Treatment Cycle 07: number analyzed (Participants) | 6
  Fatigue - Treatment Cycle 07 | 9.259 (12.989)
  Fatigue - Treatment Cycle 08: number analyzed (Participants) | 6
  Fatigue - Treatment Cycle 08 | 16.667 (18.257)
  Fatigue - Treatment Cycle 09: number analyzed (Participants) | 3
  Fatigue - Treatment Cycle 09 | 14.815 (16.973)
  Fatigue - Treatment Cycle 10: number analyzed (Participants) | 3
  Fatigue - Treatment Cycle 10 | 14.815 (16.973)
  Fatigue - Treatment Cycle 11: number analyzed (Participants) | 3
  Fatigue - Treatment Cycle 11 | 18.519 (32.075)
  Fatigue - Treatment Cycle 12: number analyzed (Participants) | 3
  Fatigue - Treatment Cycle 12 | 7.407 (23.130)
  Fatigue - Treatment Cycle 13: number analyzed (Participants) | 1
  Fatigue - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Fatigue - Treatment Cycle 14: number analyzed (Participants) | 2
  Fatigue - Treatment Cycle 14 | 0.000 (0.000)
  Fatigue - Treatment Cycle 15: number analyzed (Participants) | 2
  Fatigue - Treatment Cycle 15 | 5.556 (7.857)
  Fatigue - Follow Up: number analyzed (Participants) | 1
  Fatigue - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Fatigue - Follow Up 2: number analyzed (Participants) | 1
  Fatigue - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Fatigue - Follow Up 3: number analyzed (Participants) | 1
  Fatigue - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Nausea and Vomiting - Baseline: number analyzed (Participants) | 22
  Nausea and Vomiting - Baseline | 6.818 (15.985)
  Nausea and Vomiting - Treatment Cycle 02: number analyzed (Participants) | 20
  Nausea and Vomiting - Treatment Cycle 02 | 2.500 (9.786)
  Nausea and Vomiting - Treatment Cycle 03: number analyzed (Participants) | 16
  Nausea and Vomiting - Treatment Cycle 03 | 3.125 (12.500)
  Nausea and Vomiting - Treatment Cycle 04: number analyzed (Participants) | 12
  Nausea and Vomiting - Treatment Cycle 04 | 0.000 (7.107)
  Nausea and Vomiting - Treatment Cycle 05: number analyzed (Participants) | 8
  Nausea and Vomiting - Treatment Cycle 05 | 2.083 (5.893)
  Nausea and Vomiting - Treatment Cycle 06: number analyzed (Participants) | 8
  Nausea and Vomiting - Treatment Cycle 06 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 07: number analyzed (Participants) | 3
  Nausea and Vomiting - Treatment Cycle 07 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 08: number analyzed (Participants) | 6
  Nausea and Vomiting - Treatment Cycle 08 | 2.778 (6.804)
  Nausea and Vomiting - Treatment Cycle 09: number analyzed (Participants) | 6
  Nausea and Vomiting - Treatment Cycle 09 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 10: number analyzed (Participants) | 3
  Nausea and Vomiting - Treatment Cycle 10 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 11: number analyzed (Participants) | 3
  Nausea and Vomiting - Treatment Cycle 11 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 12: number analyzed (Participants) | 3
  Nausea and Vomiting - Treatment Cycle 12 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 13: number analyzed (Participants) | 1
  Nausea and Vomiting - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Nausea and Vomiting - Treatment Cycle 14: number analyzed (Participants) | 2
  Nausea and Vomiting - Treatment Cycle 14 | 0.000 (0.000)
  Nausea and Vomiting - Treatment Cycle 15: number analyzed (Participants) | 2
  Nausea and Vomiting - Treatment Cycle 15 | 0.000 (0.000)
  Nausea and Vomiting - Follow Up: number analyzed (Participants) | 1
  Nausea and Vomiting - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Nausea and Vomiting - Follow Up 2: number analyzed (Participants) | 1
  Nausea and Vomiting - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Nausea and Vomiting - Follow Up 3: number analyzed (Participants) | 1
  Nausea and Vomiting - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain - Baseline: number analyzed (Participants) | 22
  Pain - Baseline | 31.061 (24.286)
  Pain -Treatment Cycle 02: number analyzed (Participants) | 20
  Pain -Treatment Cycle 02 | -2.500 (23.116)
  Pain -Treatment Cycle 03: number analyzed (Participants) | 16
  Pain -Treatment Cycle 03 | -4.167 (21.517)
  Pain -Treatment Cycle 04: number analyzed (Participants) | 12
  Pain -Treatment Cycle 04 | -1.389 (18.060)
  Pain -Treatment Cycle 05: number analyzed (Participants) | 8
  Pain -Treatment Cycle 05 | 6.250 (23.465)
  Pain -Treatment Cycle 06: number analyzed (Participants) | 8
  Pain -Treatment Cycle 06 | 4.167 (24.801)
  Pain -Treatment Cycle 07: number analyzed (Participants) | 6
  Pain -Treatment Cycle 07 | 5.556 (17.213)
  Pain -Treatment Cycle 08: number analyzed (Participants) | 6
  Pain -Treatment Cycle 08 | 16.667 (29.814)
  Pain -Treatment Cycle 09: number analyzed (Participants) | 3
  Pain -Treatment Cycle 09 | 27.778 (34.694)
  Pain -Treatment Cycle 10: number analyzed (Participants) | 3
  Pain -Treatment Cycle 10 | 5.556 (9.623)
  Pain -Treatment Cycle 11: number analyzed (Participants) | 3
  Pain -Treatment Cycle 11 | 22.222 (19.245)
  Pain -Treatment Cycle 12: number analyzed (Participants) | 3
  Pain -Treatment Cycle 12 | 11.111 (19.245)
  Pain -Treatment Cycle 13: number analyzed (Participants) | 1
  Pain -Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain -Treatment Cycle 14: number analyzed (Participants) | 2
  Pain -Treatment Cycle 14 | 8.333 (11.785)
  Pain -Treatment Cycle 15: number analyzed (Participants) | 2
  Pain -Treatment Cycle 15 | 16.667 (23.570)
  Pain - Follow Up: number analyzed (Participants) | 1
  Pain - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain - Follow Up 2: number analyzed (Participants) | 1
  Pain - Follow Up 2 | -16.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain - Follow Up 3: number analyzed (Participants) | 1
  Pain - Follow Up 3 | -16.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Baseline: number analyzed (Participants) | 22
  Dyspnoea - Baseline | 25.758 (22.845)
  Dyspnoea - Treatment Cycle 02: number analyzed (Participants) | 20
  Dyspnoea - Treatment Cycle 02 | 3.333 (30.397)
  Dyspnoea - Treatment Cycle 03: number analyzed (Participants) | 16
  Dyspnoea - Treatment Cycle 03 | 6.250 (21.837)
  Dyspnoea - Treatment Cycle 04: number analyzed (Participants) | 12
  Dyspnoea - Treatment Cycle 04 | 2.778 (17.164)
  Dyspnoea - Treatment Cycle 05: number analyzed (Participants) | 8
  Dyspnoea - Treatment Cycle 05 | 8.333 (15.430)
  Dyspnoea - Treatment Cycle 06: number analyzed (Participants) | 8
  Dyspnoea - Treatment Cycle 06 | 12.500 (17.252)
  Dyspnoea - Treatment Cycle 07: number analyzed (Participants) | 6
  Dyspnoea - Treatment Cycle 07 | 5.556 (13.608)
  Dyspnoea - Treatment Cycle 08: number analyzed (Participants) | 6
  Dyspnoea - Treatment Cycle 08 | 11.111 (17.213)
  Dyspnoea - Treatment Cycle 09: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 09 | 33.333 (0.000)
  Dyspnoea - Treatment Cycle 10: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 10 | 11.111 (19.245)
  Dyspnoea - Treatment Cycle 11: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 11 | 11.111 (19.245)
  Dyspnoea - Treatment Cycle 12: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 12 | 11.111 (19.245)
  Dyspnoea - Treatment Cycle 13: number analyzed (Participants) | 1
  Dyspnoea - Treatment Cycle 13 | 33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Treatment Cycle 14: number analyzed (Participants) | 2
  Dyspnoea - Treatment Cycle 14 | 16.667 (23.570)
  Dyspnoea - Treatment Cycle 15: number analyzed (Participants) | 2
  Dyspnoea - Treatment Cycle 15 | 16.667 (23.570)
  Dyspnoea - Follow Up: number analyzed (Participants) | 1
  Dyspnoea - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Follow Up 2: number analyzed (Participants) | 1
  Dyspnoea - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Follow Up 3: number analyzed (Participants) | 1
  Dyspnoea - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Insomnia - Baseline: number analyzed (Participants) | 22
  Insomnia - Baseline | 27.273 (22.150)
  Insomnia - Treatment Cycle 02: number analyzed (Participants) | 20
  Insomnia - Treatment Cycle 02 | 5.000 (29.170)
  Insomnia - Treatment Cycle 03: number analyzed (Participants) | 16
  Insomnia - Treatment Cycle 03 | 6.250 (27.806)
  Insomnia - Treatment Cycle 04: number analyzed (Participants) | 12
  Insomnia - Treatment Cycle 04 | 0.000 (24.618)
  Insomnia - Treatment Cycle 05: number analyzed (Participants) | 8
  Insomnia - Treatment Cycle 05 | 4.167 (27.817)
  Insomnia - Treatment Cycle 06: number analyzed (Participants) | 8
  Insomnia - Treatment Cycle 06 | 8.333 (29.547)
  Insomnia - Treatment Cycle 07: number analyzed (Participants) | 6
  Insomnia - Treatment Cycle 07 | 5.556 (25.092)
  Insomnia - Treatment Cycle 08: number analyzed (Participants) | 6
  Insomnia - Treatment Cycle 08 | 0.000 (29.814)
  Insomnia - Treatment Cycle 09: number analyzed (Participants) | 3
  Insomnia - Treatment Cycle 09 | 11.111 (19.245)
  Insomnia - Treatment Cycle 10: number analyzed (Participants) | 3
  Insomnia - Treatment Cycle 10 | 11.111 (19.245)
  Insomnia - Treatment Cycle 11: number analyzed (Participants) | 3
  Insomnia - Treatment Cycle 11 | 22.222 (19.245)
  Insomnia - Treatment Cycle 12: number analyzed (Participants) | 3
  Insomnia - Treatment Cycle 12 | 11.111 (19.245)
  Insomnia - Treatment Cycle 13: number analyzed (Participants) | 1
  Insomnia - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Insomnia - Treatment Cycle 14: number analyzed (Participants) | 2
  Insomnia - Treatment Cycle 14 | 0.000 (0.000)
  Insomnia - Treatment Cycle 15: number analyzed (Participants) | 2
  Insomnia - Treatment Cycle 15 | 16.667 (23.570)
  Insomnia - Follow Up: number analyzed (Participants) | 1
  Insomnia - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Insomnia - Follow Up 2: number analyzed (Participants) | 1
  Insomnia - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Insomnia - Follow Up 3: number analyzed (Participants) | 1
  Insomnia - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Appetite Loss - Baseline: number analyzed (Participants) | 22
  Appetite Loss - Baseline | 27.273 (24.422)
  Appetite Loss - Treatment Cycle 02: number analyzed (Participants) | 20
  Appetite Loss - Treatment Cycle 02 | -1.667 (29.568)
  Appetite Loss - Treatment Cycle 03: number analyzed (Participants) | 16
  Appetite Loss - Treatment Cycle 03 | -6.250 (27.806)
  Appetite Loss - Treatment Cycle 04: number analyzed (Participants) | 12
  Appetite Loss - Treatment Cycle 04 | 2.778 (22.285)
  Appetite Loss - Treatment Cycle 05: number analyzed (Participants) | 8
  Appetite Loss - Treatment Cycle 05 | 4.167 (21.362)
  Appetite Loss - Treatment Cycle 06: number analyzed (Participants) | 8
  Appetite Loss - Treatment Cycle 06 | 4.167 (21.362)
  Appetite Loss - Treatment Cycle 07: number analyzed (Participants) | 6
  Appetite Loss - Treatment Cycle 07 | -5.556 (13.608)
  Appetite Loss - Treatment Cycle 08: number analyzed (Participants) | 6
  Appetite Loss - Treatment Cycle 08 | 0.000 (21.082)
  Appetite Loss - Treatment Cycle 09: number analyzed (Participants) | 3
  Appetite Loss - Treatment Cycle 09 | -11.111 (19.245)
  Appetite Loss - Treatment Cycle 10: number analyzed (Participants) | 3
  Appetite Loss - Treatment Cycle 10 | 0.000 (33.333)
  Appetite Loss - Treatment Cycle 11: number analyzed (Participants) | 3
  Appetite Loss - Treatment Cycle 11 | 11.111 (19.245)
  Appetite Loss - Treatment Cycle 12: number analyzed (Participants) | 3
  Appetite Loss - Treatment Cycle 12 | -11.111 (19.245)
  Appetite Loss - Treatment Cycle 13: number analyzed (Participants) | 1
  Appetite Loss - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Appetite Loss - Treatment Cycle 14: number analyzed (Participants) | 2
  Appetite Loss - Treatment Cycle 14 | 16.667 (23.570)
  Appetite Loss - Treatment Cycle 15: number analyzed (Participants) | 2
  Appetite Loss - Treatment Cycle 15 | 16.667 (23.570)
  Appetite Loss - Follow Up: number analyzed (Participants) | 1
  Appetite Loss - Follow Up | 33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Appetite Loss - Follow Up 2: number analyzed (Participants) | 1
  Appetite Loss - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Appetite Loss - Follow Up 3: number analyzed (Participants) | 1
  Appetite Loss - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Constipation - Baseline: number analyzed (Participants) | 22
  Constipation - Baseline | 15.152 (16.988)
  Constipation - Treatment Cycle 02: number analyzed (Participants) | 20
  Constipation - Treatment Cycle 02 | -3.333 (23.939)
  Constipation - Treatment Cycle 03: number analyzed (Participants) | 16
  Constipation - Treatment Cycle 03 | 6.250 (30.353)
  Constipation - Treatment Cycle 04: number analyzed (Participants) | 12
  Constipation - Treatment Cycle 04 | -5.556 (12.975)
  Constipation - Treatment Cycle 05: number analyzed (Participants) | 8
  Constipation - Treatment Cycle 05 | -4.167 (21.362)
  Constipation - Treatment Cycle 06: number analyzed (Participants) | 8
  Constipation - Treatment Cycle 06 | -8.333 (15.430)
  Constipation - Treatment Cycle 07: number analyzed (Participants) | 6
  Constipation - Treatment Cycle 07 | -5.556 (13.608)
  Constipation - Treatment Cycle 08: number analyzed (Participants) | 6
  Constipation - Treatment Cycle 08 | -5.556 (13.608)
  Constipation - Treatment Cycle 09: number analyzed (Participants) | 3
  Constipation - Treatment Cycle 09 | -11.111 (19.245)
  Constipation - Treatment Cycle 10: number analyzed (Participants) | 3
  Constipation - Treatment Cycle 10 | 0.000 (33.333)
  Constipation - Treatment Cycle 11: number analyzed (Participants) | 3
  Constipation - Treatment Cycle 11 | 11.111 (19.245)
  Constipation - Treatment Cycle 12: number analyzed (Participants) | 3
  Constipation - Treatment Cycle 12 | 0.000 (33.333)
  Constipation - Treatment Cycle 13: number analyzed (Participants) | 1
  Constipation - Treatment Cycle 13 | 33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Constipation - Treatment Cycle 14: number analyzed (Participants) | 2
  Constipation - Treatment Cycle 14 | 0.000 (0.000)
  Constipation - Treatment Cycle 15: number analyzed (Participants) | 2
  Constipation - Treatment Cycle 15 | 16.667 (23.570)
  Constipation - Follow Up: number analyzed (Participants) | 1
  Constipation - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Constipation - Follow Up 2: number analyzed (Participants) | 1
  Constipation - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Constipation - Follow Up 3: number analyzed (Participants) | 1
  Constipation - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Diarrhoea - Baseline: number analyzed (Participants) | 22
  Diarrhoea - Baseline | 9.091 (18.349)
  Diarrhoea - Treatment Cycle 02: number analyzed (Participants) | 20
  Diarrhoea - Treatment Cycle 02 | -3.333 (18.417)
  Diarrhoea - Treatment Cycle 03: number analyzed (Participants) | 16
  Diarrhoea - Treatment Cycle 03 | -4.167 (20.638)
  Diarrhoea - Treatment Cycle 04: number analyzed (Participants) | 12
  Diarrhoea - Treatment Cycle 04 | -8.333 (20.719)
  Diarrhoea - Treatment Cycle 05: number analyzed (Participants) | 8
  Diarrhoea - Treatment Cycle 05 | -4.167 (11.785)
  Diarrhoea - Treatment Cycle 06: number analyzed (Participants) | 8
  Diarrhoea - Treatment Cycle 06 | -4.167 (11.785)
  Diarrhoea - Treatment Cycle 07: number analyzed (Participants) | 6
  Diarrhoea - Treatment Cycle 07 | -5.556 (13.608)
  Diarrhoea - Treatment Cycle 08: number analyzed (Participants) | 6
  Diarrhoea - Treatment Cycle 08 | 0.000 (21.082)
  Diarrhoea - Treatment Cycle 09: number analyzed (Participants) | 3
  Diarrhoea - Treatment Cycle 09 | -11.111 (19.245)
  Diarrhoea - Treatment Cycle 10: number analyzed (Participants) | 3
  Diarrhoea - Treatment Cycle 10 | -11.111 (19.245)
  Diarrhoea - Treatment Cycle 11: number analyzed (Participants) | 3
  Diarrhoea - Treatment Cycle 11 | 0.000 (33.333)
  Diarrhoea - Treatment Cycle 12: number analyzed (Participants) | 3
  Diarrhoea - Treatment Cycle 12 | -11.111 (19.245)
  Diarrhoea - Treatment Cycle 13: number analyzed (Participants) | 1
  Diarrhoea - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Diarrhoea - Treatment Cycle 14: number analyzed (Participants) | 2
  Diarrhoea - Treatment Cycle 14 | 0.000 (0.000)
  Diarrhoea - Treatment Cycle 15: number analyzed (Participants) | 2
  Diarrhoea - Treatment Cycle 15 | 16.667 (23.570)
  Diarrhoea - Follow Up: number analyzed (Participants) | 1
  Diarrhoea - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Diarrhoea - Follow Up 2: number analyzed (Participants) | 1
  Diarrhoea - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Diarrhoea - Follow Up 3: number analyzed (Participants) | 1
  Diarrhoea - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Financial Difficulties - Baseline: number analyzed (Participants) | 22
  Financial Difficulties - Baseline | 60.606 (33.549)
  Financial Difficulties - Treatment Cycle 02: number analyzed (Participants) | 20
  Financial Difficulties - Treatment Cycle 02 | -8.333 (26.213)
  Financial Difficulties - Treatment Cycle 03: number analyzed (Participants) | 16
  Financial Difficulties - Treatment Cycle 03 | -10.417 (26.440)
  Financial Difficulties - Treatment Cycle 04: number analyzed (Participants) | 12
  Financial Difficulties - Treatment Cycle 04 | -11.111 (25.950)
  Financial Difficulties - Treatment Cycle 05: number analyzed (Participants) | 8
  Financial Difficulties - Treatment Cycle 05 | -16.667 (25.198)
  Financial Difficulties - Treatment Cycle 06: number analyzed (Participants) | 8
  Financial Difficulties - Treatment Cycle 06 | -33.333 (30.861)
  Financial Difficulties - Treatment Cycle 07: number analyzed (Participants) | 6
  Financial Difficulties - Treatment Cycle 07 | -27.778 (32.773)
  Financial Difficulties - Treatment Cycle 08: number analyzed (Participants) | 6
  Financial Difficulties - Treatment Cycle 08 | -22.222 (40.369)
  Financial Difficulties - Treatment Cycle 09: number analyzed (Participants) | 3
  Financial Difficulties - Treatment Cycle 09 | -22.222 (50.918)
  Financial Difficulties - Treatment Cycle 10: number analyzed (Participants) | 3
  Financial Difficulties - Treatment Cycle 10 | -22.222 (50.918)
  Financial Difficulties - Treatment Cycle 11: number analyzed (Participants) | 3
  Financial Difficulties - Treatment Cycle 11 | -11.111 (50.918)
  Financial Difficulties - Treatment Cycle 12: number analyzed (Participants) | 3
  Financial Difficulties - Treatment Cycle 12 | -11.111 (50.918)
  Financial Difficulties - Treatment Cycle 13: number analyzed (Participants) | 1
  Financial Difficulties - Treatment Cycle 13 | -66.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Financial Difficulties - Treatment Cycle 14: number analyzed (Participants) | 2
  Financial Difficulties - Treatment Cycle 14 | 0.000 (0.000)
  Financial Difficulties - Treatment Cycle 15: number analyzed (Participants) | 2
  Financial Difficulties - Treatment Cycle 15 | -16.667 (23.570)
  Financial Difficulties - Follow Up: number analyzed (Participants) | 1
  Financial Difficulties - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Financial Difficulties - Follow Up 2: number analyzed (Participants) | 1
  Financial Difficulties - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Financial Difficulties - Follow Up 3: number analyzed (Participants) | 1
  Financial Difficulties - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.

18. Secondary Outcome: Change From Baseline in Lung Cancer Related Symptoms
Description: The EORTC QLQ-LC13 is a specific module for lung cancer. It consists of 13 items covering lung cancer symptoms (dyspnoea, coughing, hemoptysis, pain in chest, pain in arm or shoulder and pain in other parts) and the side effects of chemo- and radiotherapy (alopecia, peripheral neuropathy, sore mouth, and dysphagia), which are divided into 10 fields, all are symptom types. All EORTC symptom scores are linearly transformed so that each score has a range of 0-100. A participant was classified as improved if a decrement of 10 points or worse was observed in the change from baseline scores. A participant was classified as worsened if a 10-point or greater increase was observed in the change from baseline scores.
Time Frame: Baseline up to approximately 1 year
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atezolizumab Plus Bevacizumab
Number analyzed (Participants) | 23
Units on a scale
  Dyspnoea - Baseline: number analyzed (Participants) | 22
  Dyspnoea - Baseline | 34.343 (20.260)
  Dyspnoea - Treatment Cycle 02: number analyzed (Participants) | 20
  Dyspnoea - Treatment Cycle 02 | -5.556 (18.557)
  Dyspnoea - Treatment Cycle 03: number analyzed (Participants) | 16
  Dyspnoea - Treatment Cycle 03 | -2.778 (20.488)
  Dyspnoea - Treatment Cycle 04: number analyzed (Participants) | 12
  Dyspnoea - Treatment Cycle 04 | -4.630 (16.723)
  Dyspnoea - Treatment Cycle 05: number analyzed (Participants) | 8
  Dyspnoea - Treatment Cycle 05 | -2.778 (19.473)
  Dyspnoea - Treatment Cycle 06: number analyzed (Participants) | 8
  Dyspnoea - Treatment Cycle 06 | 5.556 (16.798)
  Dyspnoea - Treatment Cycle 07: number analyzed (Participants) | 6
  Dyspnoea - Treatment Cycle 07 | 0.000 (14.055)
  Dyspnoea - Treatment Cycle 08: number analyzed (Participants) | 6
  Dyspnoea - Treatment Cycle 08 | 0.000 (22.222)
  Dyspnoea - Treatment Cycle 09: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 09 | 11.111 (0.000)
  Dyspnoea - Treatment Cycle 10: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 10 | 7.407 (16.973)
  Dyspnoea - Treatment Cycle 11: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 11 | 7.407 (6.415)
  Dyspnoea - Treatment Cycle 12: number analyzed (Participants) | 3
  Dyspnoea - Treatment Cycle 12 | 7.407 (16.973)
  Dyspnoea - Treatment Cycle 13: number analyzed (Participants) | 1
  Dyspnoea - Treatment Cycle 13 | 11.111 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Follow Up: number analyzed (Participants) | 1
  Dyspnoea - Follow Up | -22.222 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Follow Up 2: number analyzed (Participants) | 1
  Dyspnoea - Follow Up 2 | -22.222 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dyspnoea - Follow Up 3: number analyzed (Participants) | 1
  Dyspnoea - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Coughing - Baseline: number analyzed (Participants) | 22
  Coughing - Baseline | 37.879 (31.363)
  Coughing - Treatment Cycle 02: number analyzed (Participants) | 20
  Coughing - Treatment Cycle 02 | 1.667 (25.305)
  Coughing - Treatment Cycle 03: number analyzed (Participants) | 16
  Coughing - Treatment Cycle 03 | 10.417 (23.472)
  Coughing - Treatment Cycle 04: number analyzed (Participants) | 12
  Coughing - Treatment Cycle 04 | 0.000 (14.213)
  Coughing - Treatment Cycle 05: number analyzed (Participants) | 8
  Coughing - Treatment Cycle 05 | 4.167 (21.362)
  Coughing - Treatment Cycle 06: number analyzed (Participants) | 8
  Coughing - Treatment Cycle 06 | 16.667 (30.861)
  Coughing - Treatment Cycle 07: number analyzed (Participants) | 6
  Coughing - Treatment Cycle 07 | 0.000 (21.082)
  Coughing - Treatment Cycle 08: number analyzed (Participants) | 6
  Coughing - Treatment Cycle 08 | 11.111 (34.427)
  Coughing - Treatment Cycle 09: number analyzed (Participants) | 3
  Coughing - Treatment Cycle 09 | 0.000 (0.000)
  Coughing - Treatment Cycle 10: number analyzed (Participants) | 3
  Coughing - Treatment Cycle 10 | -11.111 (19.245)
  Coughing - Treatment Cycle 11: number analyzed (Participants) | 3
  Coughing - Treatment Cycle 11 | -11.111 (19.245)
  Coughing - Treatment Cycle 12: number analyzed (Participants) | 3
  Coughing - Treatment Cycle 12 | -11.111 (19.245)
  Coughing - Treatment Cycle 13: number analyzed (Participants) | 1
  Coughing - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Coughing - Treatment Cycle 14: number analyzed (Participants) | 2
  Coughing - Treatment Cycle 14 | 0.000 (47.140)
  Coughing - Treatment Cycle 15: number analyzed (Participants) | 2
  Coughing - Treatment Cycle 15 | 0.000 (0.00)
  Coughing - Follow Up: number analyzed (Participants) | 1
  Coughing - Follow Up | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Coughing - Follow Up 2: number analyzed (Participants) | 1
  Coughing - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Coughing - Follow Up 3: number analyzed (Participants) | 1
  Coughing - Follow Up 3 | -66.667 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Hemoptysis - Baseline | 4.545 (15.585)
  Hemoptysis - Treatment Cycle 02: number analyzed (Participants) | 20
  Hemoptysis - Treatment Cycle 02 | -1.667 (13.134)
  Hemoptysis - Treatment Cycle 03: number analyzed (Participants) | 16
  Hemoptysis - Treatment Cycle 03 | -2.083 (8.333)
  Hemoptysis - Treatment Cycle 04: number analyzed (Participants) | 12
  Hemoptysis - Treatment Cycle 04 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 05: number analyzed (Participants) | 8
  Hemoptysis - Treatment Cycle 05 | -4.167 (11.785)
  Hemoptysis - Treatment Cycle 06: number analyzed (Participants) | 8
  Hemoptysis - Treatment Cycle 06 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 07: number analyzed (Participants) | 6
  Hemoptysis - Treatment Cycle 07 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 08: number analyzed (Participants) | 6
  Hemoptysis - Treatment Cycle 08 | 11.111 (27.217)
  Hemoptysis - Treatment Cycle 09: number analyzed (Participants) | 3
  Hemoptysis - Treatment Cycle 09 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 10: number analyzed (Participants) | 3
  Hemoptysis - Treatment Cycle 10 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 11: number analyzed (Participants) | 3
  Hemoptysis - Treatment Cycle 11 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 12: number analyzed (Participants) | 3
  Hemoptysis - Treatment Cycle 12 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 13: number analyzed (Participants) | 1
  Hemoptysis - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Hemoptysis - Treatment Cycle 14: number analyzed (Participants) | 2
  Hemoptysis - Treatment Cycle 14 | 0.000 (0.000)
  Hemoptysis - Treatment Cycle 15: number analyzed (Participants) | 2
  Hemoptysis - Treatment Cycle 15 | 0.000 (0.000)
  Hemoptysis - Follow Up: number analyzed (Participants) | 1
  Hemoptysis - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Hemoptysis - Follow Up 2: number analyzed (Participants) | 1
  Hemoptysis - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Hemoptysis - Follow Up 3: number analyzed (Participants) | 1
  Hemoptysis - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Sore mouth - Baseline: number analyzed (Participants) | 22
  Sore mouth - Baseline | 3.030 (9.808)
  Sore mouth - Treatment Cycle 02: number analyzed (Participants) | 20
  Sore mouth - Treatment Cycle 02 | 6.667 (20.520)
  Sore mouth - Treatment Cycle 03: number analyzed (Participants) | 16
  Sore mouth - Treatment Cycle 03 | 4.167 (20.638)
  Sore mouth - Treatment Cycle 04: number analyzed (Participants) | 12
  Sore mouth - Treatment Cycle 04 | 0.000 (20.101)
  Sore mouth - Treatment Cycle 05: number analyzed (Participants) | 8
  Sore mouth - Treatment Cycle 05 | 4.167 (11.785)
  Sore mouth - Treatment Cycle 06: number analyzed (Participants) | 8
  Sore mouth - Treatment Cycle 06 | -4.167 (11.785)
  Sore mouth - Treatment Cycle 07: number analyzed (Participants) | 6
  Sore mouth - Treatment Cycle 07 | 5.556 (13.608)
  Sore mouth - Treatment Cycle 08: number analyzed (Participants) | 6
  Sore mouth - Treatment Cycle 08 | 5.556 (13.608)
  Sore mouth - Treatment Cycle 09: number analyzed (Participants) | 3
  Sore mouth - Treatment Cycle 09 | 0.000 (0.000)
  Sore mouth - Treatment Cycle 10: number analyzed (Participants) | 3
  Sore mouth - Treatment Cycle 10 | 0.000 (0.000)
  Sore mouth - Treatment Cycle 11: number analyzed (Participants) | 3
  Sore mouth - Treatment Cycle 11 | 0.000 (0.000)
  Sore mouth - Treatment Cycle 12: number analyzed (Participants) | 3
  Sore mouth - Treatment Cycle 12 | 0.000 (0.000)
  Sore mouth - Treatment Cycle 13: number analyzed (Participants) | 1
  Sore mouth - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Sore mouth - Treatment Cycle 14: number analyzed (Participants) | 2
  Sore mouth - Treatment Cycle 14 | 0.000 (0.000)
  Sore mouth - Treatment Cycle 15: number analyzed (Participants) | 2
  Sore mouth - Treatment Cycle 15 | 0.000 (0.000)
  Sore mouth - Follow Up: number analyzed (Participants) | 1
  Sore mouth - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Sore mouth - Follow Up 2: number analyzed (Participants) | 1
  Sore mouth - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Sore mouth - Follow Up 3: number analyzed (Participants) | 1
  Sore mouth - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dysphagia - Baseline: number analyzed (Participants) | 22
  Dysphagia - Baseline | 10.606 (15.891)
  Dysphagia - Treatment Cycle 02: number analyzed (Participants) | 20
  Dysphagia - Treatment Cycle 02 | 5.000 (24.839)
  Dysphagia - Treatment Cycle 03: number analyzed (Participants) | 16
  Dysphagia - Treatment Cycle 03 | 0.000 (12.172)
  Dysphagia - Treatment Cycle 04: number analyzed (Participants) | 12
  Dysphagia - Treatment Cycle 04 | -2.778 (9.623)
  Dysphagia - Treatment Cycle 05: number analyzed (Participants) | 8
  Dysphagia - Treatment Cycle 05 | 0.000 (0.000)
  Dysphagia - Treatment Cycle 06: number analyzed (Participants) | 8
  Dysphagia - Treatment Cycle 06 | -8.333 (15.430)
  Dysphagia - Treatment Cycle 07: number analyzed (Participants) | 6
  Dysphagia - Treatment Cycle 07 | -5.556 (13.608)
  Dysphagia - Treatment Cycle 08: number analyzed (Participants) | 6
  Dysphagia - Treatment Cycle 08 | -5.556 (13.608)
  Dysphagia - Treatment Cycle 09: number analyzed (Participants) | 3
  Dysphagia - Treatment Cycle 09 | -11.111 (19.245)
  Dysphagia - Treatment Cycle 10: number analyzed (Participants) | 3
  Dysphagia - Treatment Cycle 10 | -11.111 (19.245)
  Dysphagia - Treatment Cycle 11: number analyzed (Participants) | 3
  Dysphagia - Treatment Cycle 11 | -11.111 (19.245)
  Dysphagia - Treatment Cycle 12: number analyzed (Participants) | 3
  Dysphagia - Treatment Cycle 12 | -11.111 (19.245)
  Dysphagia - Treatment Cycle 13: number analyzed (Participants) | 1
  Dysphagia - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dysphagia - Treatment Cycle 14: number analyzed (Participants) | 2
  Dysphagia - Treatment Cycle 14 | -16.667 (23.570)
  Dysphagia - Treatment Cycle 15: number analyzed (Participants) | 2
  Dysphagia - Treatment Cycle 15 | -16.667 (23.570)
  Dysphagia - Follow Up: number analyzed (Participants) | 1
  Dysphagia - Follow Up | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dysphagia - Follow Up 2: number analyzed (Participants) | 1
  Dysphagia - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Dysphagia - Follow Up 3: number analyzed (Participants) | 1
  Dysphagia - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Peripheral neuropathy - Baseline: number analyzed (Participants) | 22
  Peripheral neuropathy - Baseline | 9.091 (18.349)
  Peripheral neuropathy - Treatment Cycle 02: number analyzed (Participants) | 20
  Peripheral neuropathy - Treatment Cycle 02 | 6.5667 (23.195)
  Peripheral neuropathy - Treatment Cycle 03: number analyzed (Participants) | 16
  Peripheral neuropathy - Treatment Cycle 03 | 4.167 (16.667)
  Peripheral neuropathy - Treatment Cycle 04: number analyzed (Participants) | 12
  Peripheral neuropathy - Treatment Cycle 04 | 8.333 (15.076)
  Peripheral neuropathy - Treatment Cycle 05: number analyzed (Participants) | 8
  Peripheral neuropathy - Treatment Cycle 05 | 12.500 (17.252)
  Peripheral neuropathy - Treatment Cycle 06: number analyzed (Participants) | 8
  Peripheral neuropathy - Treatment Cycle 06 | 12.500 (17.252)
  Peripheral neuropathy - Treatment Cycle 07: number analyzed (Participants) | 6
  Peripheral neuropathy - Treatment Cycle 07 | 11.111 (17.213)
  Peripheral neuropathy - Treatment Cycle 08: number analyzed (Participants) | 6
  Peripheral neuropathy - Treatment Cycle 08 | 11.111 (17.213)
  Peripheral neuropathy - Treatment Cycle 09: number analyzed (Participants) | 3
  Peripheral neuropathy - Treatment Cycle 09 | 0.000 (0.000)
  Peripheral neuropathy - Treatment Cycle 10: number analyzed (Participants) | 3
  Peripheral neuropathy - Treatment Cycle 10 | 0.000 (0.000)
  Peripheral neuropathy - Treatment Cycle 11: number analyzed (Participants) | 3
  Peripheral neuropathy - Treatment Cycle 11 | 11.111 (19.245)
  Peripheral neuropathy - Treatment Cycle 12: number analyzed (Participants) | 3
  Peripheral neuropathy - Treatment Cycle 12 | 0.000 (0.000)
  Peripheral neuropathy - Treatment Cycle 13: number analyzed (Participants) | 1
  Peripheral neuropathy - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Peripheral neuropathy - Treatment Cycle 14: number analyzed (Participants) | 2
  Peripheral neuropathy - Treatment Cycle 14 | 0.000 (0.000)
  Peripheral neuropathy - Treatment Cycle 15: number analyzed (Participants) | 2
  Peripheral neuropathy - Treatment Cycle 15 | 0.000 (0.000)
  Peripheral neuropathy - Follow Up: number analyzed (Participants) | 1
  Peripheral neuropathy - Follow Up | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Peripheral neuropathy - Follow Up 2: number analyzed (Participants) | 1
  Peripheral neuropathy - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Peripheral neuropathy - Follow Up 3: number analyzed (Participants) | 1
  Peripheral neuropathy - Follow Up 3 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Alopecia -Baseline: number analyzed (Participants) | 22
  Alopecia -Baseline | 16.667 (26.726)
  Alopecia - Treatment Cycle 02: number analyzed (Participants) | 20
  Alopecia - Treatment Cycle 02 | -3.333 (18.417)
  Alopecia - Treatment Cycle 03: number analyzed (Participants) | 16
  Alopecia - Treatment Cycle 03 | -12.500 (29.502)
  Alopecia - Treatment Cycle 04: number analyzed (Participants) | 12
  Alopecia - Treatment Cycle 04 | -13.889 (22.285)
  Alopecia - Treatment Cycle 05: number analyzed (Participants) | 8
  Alopecia - Treatment Cycle 05 | -8.333 (23.570)
  Alopecia - Treatment Cycle 06: number analyzed (Participants) | 8
  Alopecia - Treatment Cycle 06 | -12.500 (24.801)
  Alopecia - Treatment Cycle 07: number analyzed (Participants) | 6
  Alopecia - Treatment Cycle 07 | -5.556 (25.092)
  Alopecia - Treatment Cycle 08: number analyzed (Participants) | 6
  Alopecia - Treatment Cycle 08 | -5.556 (25.092)
  Alopecia - Treatment Cycle 09: number analyzed (Participants) | 3
  Alopecia - Treatment Cycle 09 | -11.111 (19.245)
  Alopecia - Treatment Cycle 10: number analyzed (Participants) | 3
  Alopecia - Treatment Cycle 10 | -11.111 (19.245)
  Alopecia - Treatment Cycle 11: number analyzed (Participants) | 3
  Alopecia - Treatment Cycle 11 | -11.111 (19.245)
  Alopecia - Treatment Cycle 12: number analyzed (Participants) | 3
  Alopecia - Treatment Cycle 12 | -11.111 (19.245)
  Alopecia - Treatment Cycle 13: number analyzed (Participants) | 1
  Alopecia - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Alopecia - Treatment Cycle 14: number analyzed (Participants) | 2
  Alopecia - Treatment Cycle 14 | -16.667 (23.570)
  Alopecia - Treatment Cycle 15: number analyzed (Participants) | 2
  Alopecia - Treatment Cycle 15 | -16.667 (23.570)
  Alopecia - Follow Up: number analyzed (Participants) | 1
  Alopecia - Follow Up | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Alopecia - Follow Up 2: number analyzed (Participants) | 1
  Alopecia - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Alopecia - Follow Up 3: number analyzed (Participants) | 1
  Alopecia - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in chest - Baseline: number analyzed (Participants) | 22
  Pain in chest - Baseline | 31.818 (29.951)
  Pain in chest - Treatment Cycle 02: number analyzed (Participants) | 20
  Pain in chest - Treatment Cycle 02 | 1.667 (29.568)
  Pain in chest - Treatment Cycle 03: number analyzed (Participants) | 16
  Pain in chest - Treatment Cycle 03 | 0.000 (29.814)
  Pain in chest - Treatment Cycle 04: number analyzed (Participants) | 12
  Pain in chest - Treatment Cycle 04 | 2.778 (22.285)
  Pain in chest - Treatment Cycle 05: number analyzed (Participants) | 8
  Pain in chest - Treatment Cycle 05 | 4.167 (33.034)
  Pain in chest - Treatment Cycle 06: number analyzed (Participants) | 8
  Pain in chest - Treatment Cycle 06 | 0.000 (25.198)
  Pain in chest - Treatment Cycle 07: number analyzed (Participants) | 6
  Pain in chest - Treatment Cycle 07 | 5.556 (32.773)
  Pain in chest - Treatment Cycle 08: number analyzed (Participants) | 6
  Pain in chest - Treatment Cycle 08 | -5.556 (25.092)
  Pain in chest - Treatment Cycle 09: number analyzed (Participants) | 3
  Pain in chest - Treatment Cycle 09 | -11.111 (19.245)
  Pain in chest - Treatment Cycle 10: number analyzed (Participants) | 3
  Pain in chest - Treatment Cycle 10 | -11.111 (19.245)
  Pain in chest - Treatment Cycle 11: number analyzed (Participants) | 3
  Pain in chest - Treatment Cycle 11 | -11.111 (19.245)
  Pain in chest - Treatment Cycle 12: number analyzed (Participants) | 3
  Pain in chest - Treatment Cycle 12 | -11.111 (19.245)
  Pain in chest - Treatment Cycle 13: number analyzed (Participants) | 1
  Pain in chest - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in chest - Treatment Cycle 14: number analyzed (Participants) | 2
  Pain in chest - Treatment Cycle 14 | -16.667 (23.570)
  Pain in chest - Treatment Cycle 15: number analyzed (Participants) | 2
  Pain in chest - Treatment Cycle 15 | -16.667 (23.570)
  Pain in chest - Follow Up: number analyzed (Participants) | 1
  Pain in chest - Follow Up | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in chest - Follow Up 2: number analyzed (Participants) | 1
  Pain in chest - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in chest - Follow Up 3: number analyzed (Participants) | 1
  Pain in chest - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in arm or shoulder -Baseline | 22 (27.273)
  Pain in arm or shoulder -Treatment Cycle 02: number analyzed (Participants) | 20
  Pain in arm or shoulder -Treatment Cycle 02 | -6.667 (31.715)
  Pain in arm or shoulder -Treatment Cycle 03: number analyzed (Participants) | 16
  Pain in arm or shoulder -Treatment Cycle 03 | -12.500 (36.260)
  Pain in arm or shoulder -Treatment Cycle 04: number analyzed (Participants) | 12
  Pain in arm or shoulder -Treatment Cycle 04 | -8.333 (35.176)
  Pain in arm or shoulder -Treatment Cycle 05: number analyzed (Participants) | 8
  Pain in arm or shoulder -Treatment Cycle 05 | -4.167 (45.207)
  Pain in arm or shoulder -Treatment Cycle 06: number analyzed (Participants) | 8
  Pain in arm or shoulder -Treatment Cycle 06 | -4.167 (41.547)
  Pain in arm or shoulder -Treatment Cycle 07: number analyzed (Participants) | 6
  Pain in arm or shoulder -Treatment Cycle 07 | 5.556 (25.092)
  Pain in arm or shoulder -Treatment Cycle 08: number analyzed (Participants) | 6
  Pain in arm or shoulder -Treatment Cycle 08 | 22.222 (40.369)
  Pain in arm or shoulder -Treatment Cycle 09: number analyzed (Participants) | 3
  Pain in arm or shoulder -Treatment Cycle 09 | 33.333 (57.735)
  Pain in arm or shoulder -Treatment Cycle 10: number analyzed (Participants) | 3
  Pain in arm or shoulder -Treatment Cycle 10 | 11.111 (50.918)
  Pain in arm or shoulder -Treatment Cycle 11: number analyzed (Participants) | 3
  Pain in arm or shoulder -Treatment Cycle 11 | 11.111 (50.918)
  Pain in arm or shoulder -Treatment Cycle 12: number analyzed (Participants) | 3
  Pain in arm or shoulder -Treatment Cycle 12 | 11.111 (50.918)
  Pain in arm or shoulder -Treatment Cycle 13: number analyzed (Participants) | 1
  Pain in arm or shoulder -Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in arm or shoulder -Treatment Cycle 14: number analyzed (Participants) | 2
  Pain in arm or shoulder -Treatment Cycle 14 | 50.000 (70.711)
  Pain in arm or shoulder -Treatment Cycle 15: number analyzed (Participants) | 2
  Pain in arm or shoulder -Treatment Cycle 15 | 16.667 (23.570)
  Pain in arm or shoulder - Follow Up: number analyzed (Participants) | 1
  Pain in arm or shoulder - Follow Up | 33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in arm or shoulder - Follow Up 2: number analyzed (Participants) | 1
  Pain in arm or shoulder - Follow Up 2 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in arm or shoulder - Follow Up 3: number analyzed (Participants) | 1
  Pain in arm or shoulder - Follow Up 3 | 33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in other parts - Baseline: number analyzed (Participants) | 22
  Pain in other parts - Baseline | 25.758 (28.971)
  Pain in other parts - Treatment Cycle 02: number analyzed (Participants) | 20
  Pain in other parts - Treatment Cycle 02 | -3.333 (23.939)
  Pain in other parts - Treatment Cycle 03: number analyzed (Participants) | 16
  Pain in other parts - Treatment Cycle 03 | -2.083 (22.669)
  Pain in other parts - Treatment Cycle 04: number analyzed (Participants) | 12
  Pain in other parts - Treatment Cycle 04 | 2.778 (22.285)
  Pain in other parts - Treatment Cycle 05: number analyzed (Participants) | 8
  Pain in other parts - Treatment Cycle 05 | 16.667 (25.198)
  Pain in other parts - Treatment Cycle 06: number analyzed (Participants) | 8
  Pain in other parts - Treatment Cycle 06 | -4.167 (21.362)
  Pain in other parts - Treatment Cycle 07: number analyzed (Participants) | 6
  Pain in other parts - Treatment Cycle 07 | -5.556 (25.092)
  Pain in other parts - Treatment Cycle 08: number analyzed (Participants) | 6
  Pain in other parts - Treatment Cycle 08 | 5.556 (32.773)
  Pain in other parts - Treatment Cycle 09: number analyzed (Participants) | 3
  Pain in other parts - Treatment Cycle 09 | -11.111 (19.245)
  Pain in other parts - Treatment Cycle 10: number analyzed (Participants) | 3
  Pain in other parts - Treatment Cycle 10 | -11.111 (19.245)
  Pain in other parts - Treatment Cycle 11: number analyzed (Participants) | 3
  Pain in other parts - Treatment Cycle 11 | -11.111 (19.245)
  Pain in other parts - Treatment Cycle 12: number analyzed (Participants) | 3
  Pain in other parts - Treatment Cycle 12 | -11.111 (19.245)
  Pain in other parts - Treatment Cycle 13: number analyzed (Participants) | 1
  Pain in other parts - Treatment Cycle 13 | 0.000 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in other parts - Treatment Cycle 14: number analyzed (Participants) | 2
  Pain in other parts - Treatment Cycle 14 | -16.667 (23.570)
  Pain in other parts - Treatment Cycle 15: number analyzed (Participants) | 2
  Pain in other parts - Treatment Cycle 15 | -16.667 (23.570)
  Pain in other parts - Follow Up: number analyzed (Participants) | 1
  Pain in other parts - Follow Up | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in other parts - Follow Up 2: number analyzed (Participants) | 1
  Pain in other parts - Follow Up 2 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.
  Pain in other parts - Follow Up 3: number analyzed (Participants) | 1
  Pain in other parts - Follow Up 3 | -33.333 (NA) — NA = Standard deviation couldn't be calculated from the data of one participant.

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 2.5 years
Arm/Group | Atezolizumab Plus Bevacizumab
All-Cause Mortality (participants affected / at risk) | 17/23
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab Plus Bevacizumab (N=23)
Death (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab Plus Bevacizumab (N=23)
Anaemia (Blood and lymphatic system disorders) | 5 (7)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (7)
Alanine aminotransferase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 6 (10)
Blood thyroid stimulating hormone increased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 5 (10)
Blood bilirubin increased (Investigations) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 2 (2)
Urinary occult blood positive (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Proteinuria (Renal and urinary disorders) | 7 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 6 (7)
Weight decreased (Investigations) | 5 (5)
Thyroxine free decreased (Investigations) | 2 (2)
White blood cells urine positive (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04426825/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT04426825/SAP_001.pdf